CLINICAL TRIAL: NCT01363947
Title: A Phase I, Open-Label Study of the Safety and Pharmacokinetics of Escalating Doses of DNIB0600A in Patients With Non-Small Cell Lung Cancer and Platinum-Resistant Ovarian Cancer
Brief Title: Safety and Pharmacokinetics of Escalating Doses of DNIB0600A in Participants With Non-Small Cell Lung Cancer (NSCLC) and Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNB4987g; GO27767 (Other: Hoffmann-La Roche); 2014-000527-25 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Non-Small Cell Lung Cancer, Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — lifastuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (DNIB0600A) (Experimental): Participants will receive IV infusions of DNIB0600A at doses ranging from 0.2 milligrams/kilogram (mg/kg) to 2.8 mg/kg q3w until dose-limiting toxicity (DLT) is reached, or up to 28 cycles.
  Interventions: Drug: DNIB0600A
- Expansion Cohort (DNIB0600A) (Experimental): Participants will receive 2.4 mg/kg, by IV infusion, of DNIB0600A q3w for up to 26 cycles.
  Interventions: Drug: DNIB0600A

INTERVENTIONS:
Drug: DNIB0600A — Several dose levels will be evaluated for DNIB0600A administered via IV infusion on Day 1 of each 21-day cycle until disease progression.

SUMMARY:
Study DNB4987g is a Phase I, multicenter, open label, dose-escalation study of DNIB0600A administered as a single agent by intravenous (IV) infusion every three weeks (q3w) to participants with non-squamous NSCLC or non-mucinous, platinum-resistant ovarian cancer. The study will be conducted in two cohorts: Dose-escalation cohort and Expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologic documentation of incurable, locally advanced or metastatic disease that has failed prior chemotherapy and for which no standard therapy exists, including the following: non-squamous NSCLC or non-mucinous and platinum-resistant ovarian cancer
* Availability and willingness to provide an adequate archival sample of tumor
* Measurable disease
* For fertile men or women of childbearing potential, documented willingness to use a highly effective means of contraception

Exclusion Criteria:

* Anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy within 4 weeks prior to study treatment
* Major surgical procedure within 4 weeks prior to study treatment
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including human immunodeficiency virus [HIV] and atypical mycobacterial disease, but excluding fungal infections of the nail beds)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Untreated or active central nervous system (CNS) metastases
* Requirement for supplemental oxygen to carry out activities of daily living
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Evidence of significant uncontrolled concomitant diseases, such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture
* For participants in the second NSCLC cohort expansion, not more than two prior regimens in the metastatic setting
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-06-14 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 2 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of causality.

SECONDARY OUTCOMES:
Cmax of DNIB0600A for Antibody-Conjugated Monomethyl Auristatin E (acMMAE), Total Antibody, and Unconjugated Monomethyl Auristatin E (MMAE) | Day 21
  Cmax is the peak concentration of a substance in blood serum.
Percentage of Participants with Antibody Formation to DNIB0600A | Up to approximately 84 weeks
  Serum samples will be analyzed to assess the prevalence of anti-drug antibodies (ADAs) at baseline and the incidence of post-baseline ADAs in each treatment group.
Percentage of Participants with Objective Response (OR) | Up to approximately 84 weeks
  OR is defined as a complete or partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST), v1.1. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum on study. Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered progression.
Duration of Objective Response (DOR) | Up to approximately 84 weeks
  OR is defined as a complete or partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST), v1.1. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum on study. Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered progression.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Maslyar, M.D., Study Director — Genentech, Inc.
Locations (7):
- United States (4):
  - HonorHealth Research Institute - Pima Center, Scottsdale, Arizona
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Univ of Texas SW Medical Ctr, Dallas, Texas
- Spain (3):
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid